CLINICAL TRIAL: NCT00921999
Title: Immune Responses to Varicella-Zoster Virus Vaccination and Infection
Brief Title: Immune Response to Varicella-Zoster Vaccination and Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090170; 09-I-0170
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2015-01-08

CONDITIONS: Chickenpox; Herpes Zoster
Keywords: Chickenpox; Shingles; Varicella; Zoster; Vaccine
MeSH Terms: conditions — Chickenpox; Herpes Zoster

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The common varicella-zoster virus causes both chickenpox and shingles. Both diseases cause rashes, but they can also have complications such as bacterial infections of the skin, pneumonia, or eye disease.
* By drawing and studying blood samples from people who have been infected with the varicella-zoster virus or who are receiving or have received the varicella vaccine, researchers hope to learn more about the immune system s response to the virus.

Objectives:

- To determine the immune system s response to the varicella virus, either in its existing form or given as part of a vaccine.

Eligibility:

* Individuals 18 years of age and older who have had or are receiving the varicella vaccine.
* Individuals 5 years of age and older who currently have chickenpox or shingles.

Design:

* Participants will visit the NIH Clinical Center for an initial physical examination, and will provide blood samples for evaluation.
* Researchers will determine the number of samples to be taken and the amount of blood to be drawn as needed based on the participants medical history and exposure to the varicella-zoster virus.

Investigators in this study will not be giving subjects either the chickenpox or shingles vaccine. They will only be looking at the response to the vaccine in persons who are receiving or have received the vaccine from their health care provider.

DETAILED DESCRIPTION:
Varicella-zoster virus (VZV) causes chickenpox (varicella) and shingles (zoster). Antibody is important for control of varicella as evidenced by the role of varicella immune globulin in limiting the severity of disease in immunocompromised persons. Limited information is available regarding the individual viral proteins to which antibodies are produced during primary infection with VZV or after vaccination. Furthermore, commercially available tests to determine seropositivity to VZV after vaccination have limited sensitivity, and improved assays are needed. We will obtain blood from persons with varicella, zoster, and those vaccinated with the varicella (not zoster) vaccine at the NIH Clinical Center and measure immune responses against specific viral proteins, look for virus in the blood, and in some cases measure immune responses against cellular proteins over time. Elucidation of these responses might help to develop more sensitive assays for VZV seropositivity after vaccination and determine how the varicella vaccine protects against varicella.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group I Frequent Follow-up Group (N=110)

1. 18 years of age or older
2. Patients about to receive the varicella vaccine, or were vaccinated within the last 5 days (if stored blood is available).
3. Both males and females
4. Subjects must be able to sign the consent form and be willing to comply with study procedures.
5. Subjects must be willing to have their blood samples stored.

Group II Infrequent Follow-up Group (N=30)

1. 18 years of age of older
2. Patient about to receive the varicella vaccine, or were vaccinated within the last 30 days (if stored blood is available).
3. Both males and females
4. Subjects must be able to sign the consent form and be willing to comply with study procedures.
5. Subjects must be willing to have their blood samples stored.

Group III Vaccine Recipients-Vaccinated in the Past (N=60)

1. 18 years of age or older
2. Patients were vaccinated with varicella vaccine at least 6 months previously and must provide written documentation of varicella vaccination
3. Both males and females
4. Subjects must be able to sign the consent form and be willing to comply with study procedures.
5. Subjects must be willing to have their blood samples stored.

Group IV Patients with Varicella or Zoster (N=110)

1. 5 years or older<TAB>
2. Patients presenting with varicella or zoster.
3. Both males and females
4. Subjects and/or parents/guardians must be able to sign the consent or assent form and be willing to comply with study procedures.
5. Subjects must be willing to have their blood samples stored.

EXCLUSION CRITERIA:

Study subjects will be excluded if they fulfill either of the following criteria:

1. Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or compromise patient safety (Groups I, II, IV who will be providing several blood samples)
2. History of chickenpox, zoster, or having received the zoster vaccine for patients in Groups I, II or III.
3. Patients in group I found to have a hemoglobin <11 gm/dl will be reassigned to group II or terminated from the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-06-15; Study Completion 2015-01-08

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Saiman L, LaRussa P, Steinberg SP, Zhou J, Baron K, Whittier S, Della-Latta P, Gershon AA. Persistence of immunity to varicella-zoster virus after vaccination of healthcare workers. Infect Control Hosp Epidemiol. 2001 May;22(5):279-83. doi: 10.1086/501900. PMID 11428437
- [Background] Sharrar RG, LaRussa P, Galea SA, Steinberg SP, Sweet AR, Keatley RM, Wells ME, Stephenson WP, Gershon AA. The postmarketing safety profile of varicella vaccine. Vaccine. 2000 Nov 22;19(7-8):916-23. doi: 10.1016/s0264-410x(00)00297-8. PMID 11115716
- [Background] Wasmuth EH, Miller WJ. Sensitive enzyme-linked immunosorbent assay for antibody to varicella-zoster virus using purified VZV glycoprotein antigen. J Med Virol. 1990 Nov;32(3):189-93. doi: 10.1002/jmv.1890320310. PMID 2177782
- [Derived] Cohen JI, Ali MA, Bayat A, Steinberg SP, Park H, Gershon AA, Burbelo PD. Detection of antibodies to varicella-zoster virus in recipients of the varicella vaccine by using a luciferase immunoprecipitation system assay. Clin Vaccine Immunol. 2014 Sep;21(9):1288-91. doi: 10.1128/CVI.00250-14. Epub 2014 Jul 2. PMID 24990909